CLINICAL TRIAL: NCT06732609
Title: Clinical Evaluation and Characterization of Normal Perioral Tissue With a New Advanced Videodermoscopy Method. A Pilot Study on Dental Students.
Brief Title: Perioral Tissue Evaluation With Advanced Videodermoscopy (FAV)
Acronym: FAV
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 3318
Record Dates: First submitted 2024-12-09; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Oral Mucosal Disorder
Keywords: Videodermoscopy; FAV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary aim of this study is to characterize and systematically document the key dermato-mucosal structures of the perioral region in physiological conditions. Relative to the anterior chin area (ACA), the authors have tried to identify and describe pores, fine lines or wrinkles, texture patterns, superficial desquamation, hair follicles, sebaceous glands, fine ridges, grooves, sebaceous ducts, and skin irregularities. The observed features of the vermilion border (VB) and vermilion zone (VZ) include variations in color, texture, and surface characteristics, alongside the presence of fine lines and grooves. Vascular patterns and capillary visibility were observed, with pigmentation patterns providing additional insights into structural uniformity and non-uniform areas. Shiny surfaces, pore visibility, and regional differences in sebaceous activity and texture were also highlighted, reflecting the complex variability across the vermilion zone. Additionally, novel dermatoscopic and FAV findings not previously described in the literature were introduced into the analysis based on the personal observations of the investigators. This allowed for a comprehensive evaluation of the skin characteristics, providing a detailed analysis for each anatomical zone studied.

DETAILED DESCRIPTION:
This pilot prospective observational cohort clinical study was conducted to evaluate and describe the characteristics of healthy perioral tissue in a cohort of young subjects. The study adheres to the STROBE guidelines, which ensure clear and comprehensive reporting of observational research. This study was executed in accordance with the ethical principles articulated in the Declaration of Helsinki (2014). In this study, several confounding factors were controlled through strict inclusion and exclusion criteria. Despite these measures, certain confounding factors such as age, gender, sun exposure, skin type, skincare product use, dietary habits, hydration status, stress levels, sleep patterns, physical activity, environmental exposure, genetic predisposition, and hormonal fluctuations were still present and accounted for in the analysis to ensure a rigorous interpretation of the findings.

We chose a sample of 40 participants to improve the reliability of variability estimates for key outcomes, such as perioral skin characteristics, which are essential for informing future larger-scale studies. This sample size also allows for the assessment of the methodology's feasibility across a more heterogeneous group, enhancing the generalizability of the results.

The Horus 1000VMF system used in this study consists of two lightweight probes (approximately 195 grams each) with a contact lens diameter of 2 cm. These probes are designed for dermatoscopic analysis and are equipped with two magnifications:

30x magnification, which provides a field of view (FOV) of 41.07 mm². 150x magnification, offering a FOV of 2.168 mm². The system's software allows for toggling between polarized and white light modes for enhanced observation. The focus of the images is controlled manually for precision in capturing details.

The FAV probe (Fluorescence Advanced Videodermatoscopy) enables imaging at a magnification of 500x, with a FOV of 0.092 mm². This probe utilizes a monochromatic light source with a wavelength of 405 nm to visualize layers of the skin in vivo that typically require biopsy and histological analysis.

For each patient, three anatomical areas of interest were identified and evaluated: the Anterior Chin Area (ACA), The transition zone between the ACA and the labial integument, also known as the Vermilion Border (VB), And the pigmented area of the lip, also known as the Vermilion Zone (VZ). Prior to image acquisition, the perioral region was prepared by cleaning the skin to remove any external residues, such as cosmetics or skincare products, that could affect image quality. When using the FAV mode, glycerol was applied to the skin surface to minimize light scattering and enhance image clarity. . Initially, macro images were acquired to capture a broader view of the region. Following this, a specific sequence was followed for the detailed analysis.

This sequential approach ensured a comprehensive evaluation of both surface and deeper skin structures across the different regions of interest. Once the images were captured, they were stored in the system's dedicated software for further analysis. This allowed the images to be saved and compared to future scans or used for diagnostic purposes.

The acquired dermatoscopic and FAV images were carefully reviewed by two independent investigators, both experienced in using the Horus 1000VMF system for clinical evaluations. The review process was conducted in a blinded manner, without knowledge of the patients' clinical characteristics, to avoid bias. In cases where there was a discrepancy between the two evaluators, a third evaluator was consulted to reach a consensus on the final interpretation of the images.

Others key parameters included age, sex, skin type based on Baumann's classification (Baumann, L. 2006), and Fitzpatrick's phototype (Fitzpatrick, T. B. 1988) classification were considered. Baumann's classification categorizes skin into four main types (normal, oily, dry, and combination). Fitzpatrick's classification, on the other hand, divides skin into six phototypes (I to VI) based on the skin's response to ultraviolet (UV) radiation, ranging from phototype I (very fair skin, always burns, never tans) to phototype VI (dark skin, never burns, deeply pigmented). These complementary systems provided a detailed characterization of the study population.

Descriptive statistics, such as means, medians, ranges, and relative frequencies, were employed to characterize the study participants and analyze the dermatoscopic and FAV findings.

ELIGIBILITY:
Inclusion Criteria:

* Age: Participants must be between 20 and 35 years old
* Health Status: Participants must be in good general health with no known systemic diseases (ASA I)
* Skin Condition: Participants must have clinically healthy skin in the target area, with no history of dermatological conditions such as eczema, psoriasis, or dermatitis
* Consent: Participants must provide written informed consent to participate in the study
* Non-Smoking: Participants should be non-smokers or have quit smoking for at least 12 months
* Exposure: Must not have been recently exposed to treatments affecting the skin in the area of interest (e.g., laser treatments, chemical peels, or topical medications) within the last 3 months

Exclusion Criteria:

* Dermatological Disorders: History of skin diseases (e.g., acne, psoriasis, eczema) or other skin conditions that could interfere with the assessment
* Chronic Illnesses: Presence of chronic systemic conditions (e.g., diabetes, autoimmune diseases) that may affect skin health
* Medications: Current use of medications or treatments that could alter skin characteristics (e.g., corticosteroids, retinoids, immunosuppressants)
* Allergies: Known allergies to topical products used during the examination
* Pregnancy or Lactation: Pregnant or breastfeeding individuals are excluded due to potential skin changes during these periods
* Recent Skin Procedures: Any recent dermatological procedures (e.g., laser therapy, chemical peels) performed within the last 3 months in the area of evaluation
* Excessive Sun Exposure: Individuals with recent excessive sun exposure or sunburns in the target area within the last 2 months
* Non-Compliance: Individuals unwilling or unable to comply with the study procedures

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: For the evaluation of healthy perioral tissues, the target population consisted of young, healthy individuals. The survey population specifically included students enrolled in the Dentistry and Dental Hygiene degree programs at the Catholic University of the Sacred Heart in Rome.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinical evaluation of oral mucosa disease | 8 weeks
  To observed the anterior chin area (ACA), the authors have tried to identify and describe pores, fine lines or wrinkles, texture patterns, superficial desquamation, hair follicles, sebaceous glands, fine ridges, grooves, sebaceous ducts, and skin irregularities.
Clinical evaluation of perioral mucosa | 8 weeks
  To observed the vermilion border (VB) and vermilion zone (VZ) include variations in color, texture, and surface characteristics, alongside the presence of fine lines and grooves. Vascular patterns and capillary visibility were observed, with pigmentation patterns providing additional insights into structural uniformity and non-uniform areas.
Clinical evaluation of surface and texture of oral muocsa | 8 weeks
  To observed shiny surfaces, pore visibility, and regional differences in sebaceous activity and texture were also highlighted, reflecting the complex variability across the vermilion zone.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Cordaro, MD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- UOC Clinica Odontoiatrica, Fondazione Policlinico Agostino Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fitzpatrick TB. The validity and practicality of sun-reactive skin types I through VI. Arch Dermatol. 1988 Jun;124(6):869-71. doi: 10.1001/archderm.124.6.869. No abstract available. PMID 3377516
- [Background] Browne RH. On the use of a pilot sample for sample size determination. Stat Med. 1995 Sep 15;14(17):1933-40. doi: 10.1002/sim.4780141709. PMID 8532986
- [Background] Gupta V, Sharma VK. Skin typing: Fitzpatrick grading and others. Clin Dermatol. 2019 Sep-Oct;37(5):430-436. doi: 10.1016/j.clindermatol.2019.07.010. Epub 2019 Jul 17. PMID 31896400
- [Background] Soglia S, Perez-Anker J, Lobos Guede N, Giavedoni P, Puig S, Malvehy J. Diagnostics Using Non-Invasive Technologies in Dermatological Oncology. Cancers (Basel). 2022 Nov 29;14(23):5886. doi: 10.3390/cancers14235886. PMID 36497368
- [Background] Sanlorenzo M, Vujic I, De Giorgi V, Tomasini C, Deboli T, Quaglino P, Fierro MT, Broganelli P. Fluorescence-advanced videodermatoscopy: a new method for in vivo skin evaluation. Br J Dermatol. 2017 Nov;177(5):e209-e210. doi: 10.1111/bjd.15594. Epub 2017 Oct 27. No abstract available. PMID 28421598
- [Background] Argenziano G, Soyer HP. Dermoscopy of pigmented skin lesions--a valuable tool for early diagnosis of melanoma. Lancet Oncol. 2001 Jul;2(7):443-9. doi: 10.1016/s1470-2045(00)00422-8. PMID 11905739
- [Background] Gonzalez S, Tannous Z. Real-time, in vivo confocal reflectance microscopy of basal cell carcinoma. J Am Acad Dermatol. 2002 Dec;47(6):869-74. doi: 10.1067/mjd.2002.124690. PMID 12451371
- [Background] Abati S, Bramati C, Bondi S, Lissoni A, Trimarchi M. Oral Cancer and Precancer: A Narrative Review on the Relevance of Early Diagnosis. Int J Environ Res Public Health. 2020 Dec 8;17(24):9160. doi: 10.3390/ijerph17249160. PMID 33302498